CLINICAL TRIAL: NCT00113516
Title: Phase 2 Study Of SU011248 As Consolidation Therapy In Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study Of SU011248 As Therapy In Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181057
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Paclitaxel; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: sunitinib

INTERVENTIONS:
Drug: carboplatin — AUC of 6 mg*min/mL via IV infusion every 21 days for 4 cycles as per institutional practices.
  Other Names: Paraplatin
Drug: paclitaxel — 175-225 mg/m2 via IV infusion every 21 days for 4 cycles as per institutional practices.
  Other Names: Taxol
Drug: sunitinib — 50 mg orally daily for 4 weeks followed by 2 weeks off treatment up to 1 year (after completing 1 year of treatment, pts deriving clinical benefit may continue to receive sunitinib in a separate continuation protocol).
  Other Names: SUTENT, SU011248

SUMMARY:
The purpose of this study is to find out if SU011248 (sunitinib) provides additional benefit when it is given after treatment with two chemotherapy drugs carboplatin and paclitaxel and also if sunitinib is safe for patients with locally advanced and metastatic Non Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC
* Stage IIIB (locally advanced with malignant effusion) or Stage IV disease
* No prior therapy for NSCLC
* Evidence of unidimensionally measurable disease

Exclusion Criteria:

* Previous treatment with systemic chemotherapy for lung cancer
* History of or known brain metastases
* NCI CTCAE Grade 3 hemorrhage within 4 weeks of starting study treatment
* Evidence of hemoptysis within 4 weeks of starting study treatment
* Serious acute or chronic illness or recent history of significant cardiac abnormality
* Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of EGFR and PDGFR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (20):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Burleson, Texas
  - Pfizer Investigational Site, Cleburne, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Mineral Wells, Texas
  - Pfizer Investigational Site, Weatherford, Texas
- Canada (2):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Montreal, Quebec
- France (2):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Villejuif

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181057&StudyName=A%20Study%20Of%20SU011248%20As%20Therapy%20In%20Patients%20With%20Locally%20Advanced%20Or%20Metastatic%20Non-Small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During Part 1, subjects received carboplatin plus paclitaxel 172-225 mg/m2. Those same subjects were eligible for continuation in Part 2 where they received sunitinib 50 mg. 66 subjects continued in Part 2.
Groups:
- Carboplatin Plus Paclitaxel: Carboplatin Plus Paclitaxel 172-225 mg/m2
- Sunitinib: Sunitinib 50 mg
Period: Part 1
Arm/Group | Carboplatin Plus Paclitaxel | Sunitinib
Started | 84 | 0
Completed | 0 (66 subjects continued into Part 2 of the study.) | 0
Not Completed | 84 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Death | 3 | 0
Not completed — Other | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Did Not Meet Entrance Criteria | 1 | 0
Not completed — Laboratory Abnormality | 1 | 0
Not completed — Ongoing | 1 | 0
Not completed — Missing | 65 | 0
Period: Part 2
Arm/Group | Carboplatin Plus Paclitaxel | Sunitinib
Started | 0 | 66
Completed | 0 | 0
Not Completed | 0 | 66
Not completed — Adverse Event | 0 | 16
Not completed — Death | 0 | 5
Not completed — Lack of Efficacy | 0 | 37
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 0 | 3
Not completed — Laboratory Abnormality | 0 | 1
Not completed — Ongoing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- First Carboplatin Plus Paclitaxel, Then Sunitinib: Part 1 = Carboplatin plus Paclitaxel 172-225 mg/m2. Part 2 = Sunitinib 50 mg
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
Age, Customized [Number; unit: participants]
  < 65 years | 53
  > = 65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Surviving at One Year
Description: Proportion of those surviving at the end of one year from the first dose of study treatment. In the absence of confirmation of death, survival time was censored at the last date the subject was known to be alive. Patients lacking data beyond the day of first dose had their survival time censored at Day 1 of treatment.
Time Frame: From start of treatment until 1 year or death
Population: Intent-to-treat (ITT) population = all subjects enrolled in the study who received at least 1 dose of paclitaxel/carboplatin.
Measure: Number; unit: proportion
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
proportion | 0.405
Statistical Analysis 1: Comparison: First Carboplatin Plus Paclitaxel, Then Sunitinib; The study was designed to test the null hypothesis that the true one-year probability of survival is 0.40 versus the alternative hypothesis that the true one-year probability of survival is at least 0.55. The sample size was determined using a One-Sample Survival design, assuming alpha=0.05 (1-sided), power= 0.90, 6 month accrual, a minimum follow-up period of 12 months, and an expectation that approximately 5% of subjects may be lost to follow-up; Test type: Superiority or Other; Kaplan-Meier; probability = 0.405, 90% CI 2-sided [0.315 to 0.494] — The probability of survival along with the corresponding confidence interval (CI) (for the log [-log (1-year survival rate)]) was calculated using a normal approximation and then back transformed to give a CI for the 1-year survival rate itself

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from start of study treatment to first documentation of objective disease progression or to death on study due to any cause, whichever was first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date - first paclitaxel/carboplatin dose date +1)/7.02.
Time Frame: From start of treatment until Day 21 of Cycles 2 and 4 (Carboplatin plus Paclitaxel), Day 28 of Cycles 1, 2, 3, 4, and even cycles thereafter (Sunitinib) or death
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
weeks | 23.1 [21.4 to 28.2]

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from start of study treatment to first documentation of objective disease progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date - first paclitaxel/carboplatin dose date +1)/7.02.
Time Frame: From start of treatment until Day 21 of Cycles 2 and 4 (Carboplatin plus Paclitaxel), Day 28 of Cycles 1, 2, 3, 4, and even cycles thereafter (Sunitinib)
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
weeks | 23.6 [22.6 to 29.3]

4. Secondary Outcome: Duration of Response (DR)
Description: DR=time from the first documentation of objective tumor response (complete response [CR] or partial response [PR]) that was subsequently confirmed to first documentation of objective disease progression or death due to any cause, whichever was first. CR=disappearance of all target lesions. PR=a > = 30% decrease in sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions. If tumor progression data included more than 1 date, first date was used. DR (in weeks) was calculated as (the end date for DR - first CR or PR that was subsequently confirmed +1)/7.02.
Time Frame: as for outcome 2
Population: ITT. DR was calculated for the subgroup of subjects with objective response. 23 subjects reported CR or PR response and were analyzed for DR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 23
weeks | 27.3 [16.3 to 40.1]

5. Secondary Outcome: Number of Subjects With Overall Confirmed Objective Disease Response
Description: Objective disease response = subjects with confirmed CR or PR according to the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.0). A CR was defined as the disappearance of all target lesions. A PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: as for outcome 3
Population: ITT
Measure: Number; unit: participants
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
participants | 23
Statistical Analysis 1: Comparison: First Carboplatin Plus Paclitaxel, Then Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 27.4, 95% CI 2-sided [18.2 to 38.2]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of study treatment to death due to any cause. OS (in months) was calculated as (date of death - date of paclitaxel/carboplatin first dose +1)/30.4. For subjects not expiring, their survival times were censored at the last date of known contact they were known to be alive. Subjects lacking data beyond the day of first dose of paclitaxel/carboplatin had their survival time censored at Day 1 of paclitaxel/carboplatin treatment.
Time Frame: From start of study treatment until death
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
months | 10.4 [8.1 to 12.2]

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Sunitinib
Description: Ctrough = the plasma concentration prior to study drug administration. On Day 28, this parameter provided and idea of the concentration at steady state since no big fluctuation was expected in a 24 hour interval.
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: Pharmacokinetic (PK) = all subjects enrolled in the study who received at least 1 dose of carboplatin/paclitaxel or sunitinib. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Groups:
- Sunitinib: Part 2 = Sunitinib 50 mg
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
nanograms (ng)/milliliter (mL)
  Cycle 1, Day 28 (n=51) | 57.69 (29.37)
  Cycle 2, Day 28 (n=36) | 50.88 (33.67)
  Cycle 3, Day 28 (n=16) | 41.55 (24.28)
  Cycle 5, Day 28 (n=6) | 38.57 (21.83)

8. Secondary Outcome: Ctrough of SU-012662 (Sunitinib's Metabolite)
Description: as for outcome 7
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: PK. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
ng/mL
  Cycle 1, Day 28 (n=51) | 27.54 (15.10)
  Cycle 2, Day 28 (n=36) | 23.47 (20.99)
  Cycle 3, Day 28 (n=16) | 18.37 (9.05)
  Cycle 5, Day 28 (n=6) | 15.67 (7.12)

9. Secondary Outcome: Ctrough of Total Drug (Sunitinib + SU-012662)
Description: as for outcome 7
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: PK. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
ng/mL
  Cycle 1, Day 28 (n=51) | 85.23 (42.22)
  Cycle 2, Day 28 (n=36) | 74.35 (51.60)
  Cycle 3, Day 28 (n=16) | 59.92 (30.72)
  Cycle 5, Day 28 (n=6) | 54.24 (27.90)

10. Secondary Outcome: Dose-Corrected Ctrough of Sunitinib
Description: Ctrough = the plasma concentration prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. This was determined due to potential dose changes throughout the study in different subjects. It was calculated as the observed values multiplied by the reference dose (50 mg) divided by the actual dose. For dose-corrected trough concentration, only trough concentration values from subjects who received sunitinib during at least the last 10 consecutive days of dosing at the same dose level were included.
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: PK. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
ng/mL
  Cycle 1, Day 28 (n=39) | 64.10 (26.84)
  Cycle 2, Day 28 (n=28) | 59.85 (40.45)
  Cycle 3, Day 28 (n=13) | 49.59 (21.86)
  Cycle 5, Day 28 (n=5) | 54.51 (13.67)

11. Secondary Outcome: Dose-Corrected Ctrough of SU-012662 (Sunitinib's Metabolite)
Description: as for outcome 10
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: PK. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
ng/mL
  Cycle 1, Day 28 (n=39) | 27.90 (14.66)
  Cycle 2, Day 28 (n=28) | 27.37 (30.55)
  Cycle 3, Day 28 (n=13) | 20.64 (9.97)
  Cycle 5, Day 28 (n=5) | 22.29 (8.35)

12. Secondary Outcome: Dose-Corrected Ctrough of Total Drug (Sunitinib + SU-012662)
Description: as for outcome 10
Time Frame: predose on Day 28 of Cycles 1, 2, 3, and 5 of Part 2
Population: PK. Subjects with plasma values below limit of quantification were excluded.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 66
ng/mL
  Cycle 1, Day 28 (n=39) | 92.00 (40.31)
  Cycle 2, Day 28 (n=28) | 87.22 (68.28)
  Cycle 3, Day 28 (n=13) | 70.24 (28.71)
  Cycle 5, Day 28 (n=5) | 76.80 (20.13)

13. Secondary Outcome: Vascular Endothelial Growth Factor Receptor 3 (VEGFR3) Concentration at Baseline
Description: Concentration of VEGFR3 at baseline.
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: Modified ITT population (MITT) = all subjects enrolled in the study who received at least 1 dose of paclitaxel/carboplatin and at least 1 dose of Sunitinib.
Measure: Mean (Standard Deviation); unit: picograms (pg)/milliliter (mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 60
picograms (pg)/milliliter (mL) | 30382.83 (19134.12)

14. Secondary Outcome: VEGFR3 Ratio to Baseline at Each Time Point
Description: VEGFR3 concentration at each time point divided by VEGFR3 concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers at baseline and at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 46
ratio
  Cycle 1, Day 28 (n=46) | 0.39 (0.201)
  Cycle 2, Day 1 (n=40) | 0.74 (0.255)
  Cycle 2, Day 28 (n=29) | 0.36 (0.165)
  Cycle 3, Day 1 (n=21) | 0.70 (0.288)
  Cycle 3, Day 28 (n=12) | 0.31 (0.111)
  Cycle 5, Day 28 (n=4) | 0.31 (0.163)

15. Secondary Outcome: VEGF-C Concentration at Baseline
Description: Concentration of VEGF-C at baseline.
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: MITT. Number of participants analyzed = number of subjects with VEGF-C data at Baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
pg/mL | 793.19 (323.770)

16. Secondary Outcome: VEGF-C Ratio to Baseline at Each Time Point
Description: VEGF-C concentration at each time point divided by VEGF-C concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers at baseline and at the specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 46
ratio
  Cycle 1, Day 28 (n=46) | 0.81 (0.342)
  Cycle 2, Day 1 (n=39) | 0.90 (0.396)
  Cycle 2, Day 28 (n=30) | 0.91 (0.577)
  Cycle 3, Day 1 (n=20) | 1.00 (0.460)
  Cycle 3, Day 28 (n=12) | 0.91 (0.340)
  Cycle 5, Day 28 (n=4) | 0.89 (0.269)

17. Secondary Outcome: Soluble E-Selectin at Baseline
Description: Concentration of soluble E-Selectin at baseline.
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: MITT. Number of participants analyzed = number of subjects with soluble E-Selectin data at Baseline.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 53
nanograms (ng)/mL | 27.06 (11.474)

18. Secondary Outcome: Soluble E-Selectin Ratio to Baseline at Each Time Point
Description: Soluble E-Selectin concentration at each time point divided by soluble E-Selectin concentration at baseline (ratio to baseline).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 4 (Day 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers at baseline and at the specified time point. At Cycle 4, Day 28, median and/or standard deviation were not able to be estimated.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 34
ratio
  Cycle 1, Day 28 (n=34) | 0.83 (0.222)
  Cycle 2, Day 1 (n=29) | 0.89 (0.287)
  Cycle 2, Day 28 (n=22) | 0.77 (0.246)
  Cycle 3, Day 1 (n=16) | 0.81 (0.224)
  Cycle 3, Day 28 (n=8) | 0.69 (0.126)
  Cycle 5, Day 28 (n=3) | 0.76 (0.354)

19. Secondary Outcome: VEGFR3 at Baseline Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median concentration of VEGFR3 at baseline stratified by tumor response (CR or PR or [SD > = 6 Weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a nonparametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 45
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=21) | 21660.00
  Cycle 1, Day 1 (PD, n=24) | 27740.00
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; p = 0.474, Wilcoxon Rank Sum Test

20. Secondary Outcome: VEGFR3 Ratio to Baseline at Each Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median VEGFR3 concentration at each time point divided by median VEGFR3 concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR or [SD > = 6 weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers at baseline and at the specified time point. No subjects had PD at Cycle 5, Day 28.
Measure: Number; unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
ratio
  Cycle 1, Day 28 (CR or PR or SD, n=16) | 0.34
  Cycle 1, Day 28 (PD, n=20) | 0.35
  Cycle 2, Day 1 (CR or PR or SD, n=19) | 0.75
  Cycle 2, Day 1 (PD, n=16) | 0.84
  Cycle 2, Day 28 (CR or PR or SD, n=15) | 0.32
  Cycle 2, Day 28 (PD, n=12) | 0.38
  Cycle 3, Day 1 (CR or PR or SD, n=15) | 0.57
  Cycle 3, Day 1 (PD, n=5) | 0.92
  Cycle 3, Day 28 (CR or PR or SD, n=11) | 0.38
  Cycle 3, Day 28 (pd, n=1) | 0.43
  Cycle 5, Day 28 (CR or PR or SD, n=4) | 0.30
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.836, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.071, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.393, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.029, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.247, Wilcoxon Rank Sum Test

21. Secondary Outcome: VEGF-C at Baseline Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median concentration of VEGF-C at baseline stratified by tumor response (CR or PR or [SD > = 6 Weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a nonparametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 44
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=20) | 704.80
  Cycle 1, Day 1 (PD, n=24) | 766.45
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; p = 0.305, Wilcoxon Rank Sum Test

22. Secondary Outcome: VEGF-C Ratio to Baseline at Each Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median VEGF-C concentration at each time point divided by median VEGF-C concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR or [SD > = 6 weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. No subjects had PD at Cycle 5, Day 28.
Measure: Number; unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
ratio
  Cycle 1, Day 28 (CR or PR or SD, n=16) | 0.73
  Cycle 1, Day 28 (PD, n=20) | 0.81
  Cycle 2, Day 1 (CR or PR or SD, n=18) | 0.87
  Cycle 2, Day 1 (PD, n=16) | 0.85
  Cycle 2, Day 28 (CR or PR or SD, n=16) | 0.89
  Cycle 2, Day 28 (PD, n=12) | 0.69
  Cycle 3, Day 1 (CR or PR or SD, n=14) | 0.89
  Cycle 3, Day 1 (PD, n=5) | 0.78
  Cycle 3, Day 28 (CR or PR or SD, n=11) | 0.85
  Cycle 3, Day 28 (PD, n=1) | 0.90
  Cycle 5, Day 28 (CR or PR or SD, n=4) | 0.78
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.738, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.438, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.236, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.287, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.772, Wilcoxon Rank Sum Test

23. Secondary Outcome: Soluble E-Selectin at Baseline Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median concentration of soluble E-selectin at baseline stratified by tumor response (CR or PR or [SD > = 6 Weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a nonparametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline (Cycle 1, Day 1) of Part 2
Population: MITT. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Number; unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 38
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=17) | 26.40
  Cycle 1, Day 1 (PD, n=21) | 27.40
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; p = 0.537, Wilcoxon Rank Sum Test

24. Secondary Outcome: Soluble E-Selectin Ratio to Baseline at Each Time Point Stratified by Tumor Response (CR or PR or [SD > = 6 Weeks] or PD)
Description: Median soluble E-selectin concentration at each time point divided by median soluble E-selectin concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR or [SD > = 6 weeks] or PD). A measure of dispersion is not included because the Wilcoxon rank sum test is a non-parametric test that makes no assumptions about the distribution of the data (eg, normality).
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 4 (Day 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. No subjects had PD at Cycle 4, Day 28 and Cycle 5, Day 28.
Measure: Number; unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 26
ratio
  Cycle 1, Day 28 (CR or PR or SD, n=10) | 0.84
  Cycle 1, Day 28 (PD, n=16) | 0.84
  Cycle 2, Day 1 (CR or PR or SD, n=13) | 0.84
  Cycle 2, Day 1 (PD, n=12) | 0.76
  Cycle 2, Day 28 (CR or PR or SD, n=10) | 0.86
  Cycle 2, Day 28 (PD, n=10) | 0.64
  Cycle 3, Day 1 (CR or PR or SD, n=10) | 0.74
  Cycle 3, Day 1 (PD, n=5) | 0.77
  Cycle 3, Day 28 (CR or PR or SD, n=7) | 0.67
  Cycle 3, Day 28 (PD, n=1) | 0.78
  Cycle 4, Day 28 (CR or PR or SD, n=1) | 1.13
  Cycle 5, Day 28 (CR or PR or SD, n=3) | 0.64
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.813, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.849, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.121, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.582, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.383, Wilcoxon Rank Sum Test

25. Secondary Outcome: Comparison of Kaplan-Meier PFS Curves After Stratification by < or > = Median Levels of VEGFR3 at Baseline and Changes From Baseline
Description: PFS = time from start of study treatment to first documentation of objective disease progression or to death on study due to any cause, whichever was first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date minus first sunitinib dose date +1)divided by 7.02. Groups are defined by < or > = median levels of VEGFR3 at Baseline and after Stratification by < or > = median changes from Baseline in VEGFR3 at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 28 (< median cutpoint) and Cycle 5, Day 28 (> = median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 60
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=30) | 13.1 [10.11 to 32.91]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 10.3 [9.12 to 16.10]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 15.8 [9.97 to 32.91]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 10.3 [6.84 to 16.81]
  Cycle 2, Day 1 (< Median Cutpoint, n=20) | 22.5 [15.81 to 33.90]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 11.1 [10.83 to 16.81]
  Cycle 2, Day 28 (< Median Cutpoint, n=14) | 16.8 [10.83 to 32.91]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 16.1 [10.97 to 33.90]
  Cycle 3, Day 1 (< Median Cutpoint, n=10) | 32.9 [22.51 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint, n=11) | 16.1 [9.97 to 33.90]
  Cycle 3, Day 28 (> = Median Cutpoint, n=6) | 32.9 [21.79 to 45.73]
  Cycle 5, Day 28 (< Median Cutpoint, n=2) | 38.3 [30.77 to 45.87]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.6782, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.61 to 2.15] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.1980, Log Rank; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.77 to 3.30] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.1344, Log Rank; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [0.82 to 3.98] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.4809, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.56 to 3.39] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.0153, Log Rank; Hazard Ratio (HR) = 3.6, 95% CI 2-sided [1.19 to 11.13] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.2085, Log Rank; Hazard Ratio (HR) = 2.7, 95% CI 2-sided [0.52 to 14.37] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 7: Comparison: Sunitinib; Cycle 5, Day 28; Test type: Superiority or Other; p = 0.8084, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.08 to 23.57] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

26. Secondary Outcome: Comparison of Kaplan-Meier PFS Curves After Stratification by < or > = Median Levels of VEGF-C at Baseline and Changes From Baseline
Description: PFS = time from start of study treatment to first documentation of objective disease progression or to death on study due to any cause, whichever was first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date minus first sunitinib dose date +1) divided by 7.02. Groups are defined by < or > = median levels of VEGF-C at Baseline and after stratification by < or > = median changes from Baseline in VEGF-C at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 28 (< median cutpoint) and Cycle 5, Day 28 (< median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=29) | 16.1 [10.97 to 32.91]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 10.1 [8.97 to 15.81]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 12.4 [8.97 to 43.30]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 11.0 [9.97 to 16.81]
  Cycle 2, Day 1 (< Median Cutpoint, n=19) | 13.1 [10.11 to 22.51]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 16.1 [10.97 to 33.90]
  Cycle 2, Day 28 (< Median Cutpoint, n=15) | 10.8 [10.11 to 16.81]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 31.8 [16.10 to 45.73]
  Cycle 3, Day 1 (< Median Cutpoint, n=10) | 19.7 [10.11 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint, n=10) | 30.8 [15.81 to 33.90]
  Cycle 3, Day 28 (> = Median Cutpoint, n=6) | 32.9 [30.77 to 45.73]
  Cycle 5, Day 28 (> = Median Cutpoint, n=2) | 37.0 [30.77 to 43.30]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.5070, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.65 to 2.39] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.4474, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.63 to 2.82] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.7599, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.40 to 1.95] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.0109, Log Rank; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.12 to 0.80] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.6878, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.43 to 3.58] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.4637, Log Rank; Hazard Ratio (HR) = 1.7, 95% CI 2-sided [0.38 to 8.12] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

27. Secondary Outcome: Comparison of Kaplan-Meier PFS Curves After Stratification by < or > = Median Levels of Soluble E-Selectin at Baseline and Changes From Baseline
Description: PFS = time from start of study treatment to first documentation of objective disease progression or to death on study due to any cause, whichever was first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date minus first sunitinib dose date +1) divided by 7.02. Groups are defined by < or > = median levels of soluble E-selectin at Baseline and after stratification by < or > = median changes from Baseline in soluble E-selectin at each time point.
Time Frame: [Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 4 (Day 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 2, Day 28 (> = median cutpoint), Cycle 3, Day 28 (< median cutpoint), and Cycles 4 and 5, Day 28 (< median cutpoint, > = median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 53
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=26) | 11.1 [9.12 to 22.51]
  Cycle 1, Day 1 (> = Median Cutpoint, n=27) | 11.0 [9.97 to 21.79]
  Cycle 1, Day 28 (< Median Cutpoint, n=17) | 11.0 [9.26 to 21.79]
  Cycle 1, Day 28 (> = Median Cutpoint, n=17) | 10.1 [6.84 to 16.10]
  Cycle 2, Day 1 (< Median Cutpoint, n=14) | 11.0 [10.11 to 45.87]
  Cycle 2, Day 1 (> = Median Cutpoint, n=15) | 16.1 [10.11 to 33.90]
  Cycle 2, Day 28 (< Median Cutpoint, n=11) | 11.0 [10.11 to 16.81]
  Cycle 3, Day 1 (< Median Cutpoint, n=8) | 33.8 [9.97 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint, n=8) | 22.5 [10.11 to 43.30]
  Cycle 3, Day 28 (> = Median Cutpoint, n=4) | 43.3 [16.10 to 43.30]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.5277, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.39 to 1.62] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.4660, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.58 to 3.29] — HR was based upon the ratio of >=Median Cutpoint group hazard to <Median Cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.5337, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.52 to 3.44] — HR was based upon the ratio of >=Median Cutpoint group hazard to <Median Cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.0712, Log Rank; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.13 to 1.13] — HR was based upon the ratio of >=Median Cutpoint group hazard to <Median Cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.2948, Log Rank; Hazard Ratio (HR) = 2.0, 95% CI 2-sided [0.54 to 7.07] — HR was based upon the ratio of >=Median Cutpoint group hazard to <Median Cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.3200, Log Rank; Hazard Ratio (HR) = 3.3, 95% CI 2-sided [0.28 to 38.48] — HR was based upon the ratio of >=Median Cutpoint group hazard to <Median Cutpoint group

28. Secondary Outcome: Comparison of Kaplan-Meier TTP Curves After Stratification by < or > = Median Levels of VEGFR3 at Baseline and Changes From Baseline
Description: TTP = time from start of study treatment to first documentation of objective disease progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first sunitinib dose date +1) divided by 7.02. Groups are defined by < or > = median levels of VEGFR3 at Baseline and after stratification by < or > = median changes from baseline in VEGFR3 at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 60
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=30) | 15.8 [10.83 to 32.91]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 11.0 [9.26 to 21.79]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 15.8 [9.97 to 32.91]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 12.4 [9.97 to 16.81]
  Cycle 2, Day 1 (< Median Cutpoint, n=20) | 30.8 [15.81 to 33.90]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 11.1 [10.83 to 16.81]
  Cycle 2, Day 28 (< Median Cutpoint, n=14) | 16.8 [10.83 to 32.91]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 16.1 [10.97 to 33.90]
  Cycle 3, Day 1 (< Median Cutpoint, n=10) | 32.9 [30.77 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint, n=11) | 16.1 [9.97 to 33.90]
  Cycle 3, Day 28 (> = Median Cutpoint, n=6) | 32.9 [21.79 to 45.73]
  Cycle 5, Day 28 (< Median Cutpoint, n=2) | 38.3 [30.77 to 45.87]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.7824, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.56 to 2.17] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.1918, Log Rank; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.77 to 3.47] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.1093, Log Rank; Hazard Ratio (HR) = 1.9, 95% CI 2-sided [0.85 to 4.30] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.4809, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.56 to 3.39] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.0110, Log Rank; Hazard Ratio (HR) = 4.2, 95% CI 2-sided [1.26 to 13.85] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.2085, Log Rank; Hazard Ratio (HR) = 2.7, 95% CI 2-sided [0.52 to 14.37] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 7: Comparison: Sunitinib; Cycle 5, Day 28; Test type: Superiority or Other; p = 0.8084, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.08 to 23.57] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

29. Secondary Outcome: Comparison of Kaplan-Meier TTP Curves After Stratification by < or > = Median Levels of VEGF-C at Baseline and Changes From Baseline
Description: TTP = time from start of study treatment to first documentation of objective disease progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first sunitinib dose date +1) divided by 7.02. Groups are defined by < or > = median levels of VEGF-C at Baseline and after stratification by < or > = median changes from Baseline in VEGF-C at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 28 (< median cutpoint), and Cycle 5, Day 28 (< median cutpoint, > = median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=29) | 16.1 [10.97 to 32.91]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 10.3 [9.26 to 16.81]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 15.8 [9.12 to 43.30]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 11.0 [9.97 to 16.81]
  Cycle 2, Day 1 (< Median Cutpoint, n=19) | 13.1 [10.11 to 16.81]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 16.1 [10.97 to 33.90]
  Cycle 2, Day 28 (< Median Cutpoint, n=15) | 10.8 [10.11 to 16.81]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 31.8 [16.10 to 45.73]
  Cycle 3, Day 1 (< Median Cutpoint, n=10) | 16.8 [10.11 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint, n=10) | 30.8 [15.81 to 33.90]
  Cycle 3, Day 28 (> = Median Cutpoint, n=6) | 32.9 [30.77 to 45.73]
  Cycle 5, Day 28 (> = Median Cutpoint, n=2) | 37.0 [30.77 to 43.30]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.5215, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.62 to 2.53] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.2504, Log Rank; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.72 to 3.49] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.8766, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.42 to 2.11] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.0109, Log Rank; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.12 to 0.80] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.5627, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.46 to 4.18] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.4637, Log Rank; Hazard Ratio (HR) = 1.7, 95% CI 2-sided [0.38 to 8.12] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

30. Secondary Outcome: Comparison of Kaplan-Meier TTP Curves After Stratification by < or > = Median Levels of Soluble E-Selectin at Baseline Changes From Baseline
Description: TTP = time from start of study treatment to first documentation of objective disease progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first sunitinib dose date +1) divided by 7.02. Groups are defined by < or > = median levels of soluble E-selectin at Baseline and after stratification by < or > = median changes from Baseline in soluble E-selectin at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 4 (Day 28), Cycle 5 (Day 28) of Part 2
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 53
weeks
  Cycle 1, Day 1 (< Median Cutpoint, n=26) | 11.1 [9.97 to 43.30]
  Cycle 1, Day 1 (> = Median Cutpoint, n=27) | 12.4 [10.11 to 33.90]
  Cycle 1, Day 28 (< Median Cutpoint, n=17) | 11.0 [9.26 to 21.79]
  Cycle 1, Day 28 (> = Median Cutpoint, n=17) | 10.1 [9.12 to 43.30]
  Cycle 2, Day 1 (< Median Cutpoint, n=14) | 11.0 [10.11 to 45.87]
  Cycle 2, Day 1 (> = Median Cutpoint, n=15) | 16.1 [10.11 to 33.90]
  Cycle 2, Day 28 (< Median Cutpoint, n=11) | 11.0 [10.11 to 16.81]
  Cycle 3, Day 1 (< Median Cutpoint, n=8) | 33.8 [9.97 to 45.87]
  Cycle 3, Day 1 (> = Median Cutpoint n=8) | 33.9 [10.11 to 43.30]
  Cycle 3, Day 28 (> = Median Cutpoint, n=4) | 43.3 [16.10 to 43.30]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.6682, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.39 to 1.84] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.6854, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.49 to 3.00] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.6028, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.49 to 3.37] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.0712, Log Rank; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.13 to 1.13] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.3411, Log Rank; Hazard Ratio (HR) = 1.9, 95% CI 2-sided [0.50 to 7.15] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.3200, Log Rank; Hazard Ratio (HR) = 3.3, 95% CI 2-sided [0.28 to 38.48] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

31. Secondary Outcome: Comparison of Kaplan-Meier OS Curves After Stratification by < or > = Median Levels of VEGFR3 at Baseline Changes From Baseline
Description: OS = time from start of study treatment to death due to any cause. OS (in months) was calculated as (date of death minus date of sunitinib first dose +1)divided by 30.4. For subjects not expiring, their survival times were censored at the last date of known contact they were known to be alive. Subjects lacking data beyond the day of first dose of sunitinib had their survival time censored at Day 1 of sunitinib treatment. Groups are defined by < or > = median levels of VEGFR3 at Baseline and after stratification by < or > = median changes from Baseline in VEGFR3 at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 1 (< median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 60
months
  Cycle 1, Day 1 (< Median Cutpoint, n=30) | 8.7 [6.55 to 20.53]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 6.1 [4.51 to 9.67]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 14.7 [5.23 to 22.89]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 7.1 [4.41 to 11.15]
  Cycle 2, Day 1 (< Median Cutpoint, n=20) | 13.7 [6.12 to 22.89]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 8.8 [6.55 to 24.47]
  Cycle 2, Day 28 (< Median Cutpoint, n=14) | 11.2 [7.11 to 22.89]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 13.3 [8.82 to 26.09]
  Cycle 3, Day 1 (> = Median Cutpoint, n=11) | 7.4 [5.07 to 13.26]
  Cycle 3, Day 28 (< Median Cutpoint, n=6) | 17.7 [13.65 to 22.89]
  Cycle 5, Day 28 (< Median Cutpoint, n=2) | 17.1 [13.65 to 20.53]
  Cycle 5, Day 28 (> = Median Cutpoint, n=2) | 13.8 [12.66 to 14.84]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.4768, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.70 to 2.17] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.1484, Log Rank; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.84 to 3.13] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.8957, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.50 to 2.18] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.5681, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.33 to 1.85] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.0074, Log Rank; Hazard Ratio (HR) = 3.8, 95% CI 2-sided [1.35 to 10.88] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.1637, Log Rank; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.06 to 1.70] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 7: Comparison: Sunitinib; Cycle 5, Day 28; Test type: Superiority or Other; p = 0.4328, Log Rank; Hazard Ratio (HR) = 2.6, 95% CI 2-sided [0.23 to 29.12] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

32. Secondary Outcome: Comparison of Kaplan-Meier OS Curves After Stratification by < or > = Median Levels of VEGF-C at Baseline and Changes From Baseline
Description: OS = time from start of study treatment to death due to any cause. OS (in months) was calculated as (date of death minus date of sunitinib first dose +1) divided by 30.4. For subjects not expiring, their survival times were censored at the last date of known contact they were known to be alive. Subjects lacking data beyond the day of first dose of sunitinib had their survival time censored at Day 1 of sunitinib treatment. Groups are defined by < or > = median levels of VEGF-C at Baseline and after stratification by < or > = median changes from Baseline in VEGF-C at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 28 (> = median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
months
  Cycle 1, Day 1 (< Median Cutpoint, n=29) | 8.5 [6.32 to 15.76]
  Cycle 1, Day 1 (> = Median Cutpoint, n=30) | 5.2 [4.41 to 12.66]
  Cycle 1, Day 28 (< Median Cutpoint, n=23) | 8.5 [5.07 to 14.84]
  Cycle 1, Day 28 (> = Median Cutpoint, n=23) | 8.8 [4.41 to 20.53]
  Cycle 2, Day 1 (< Median Cutpoint, n=19) | 9.7 [5.20 to 14.84]
  Cycle 2, Day 1 (> = Median Cutpoint, n=20) | 12.7 [6.55 to 22.89]
  Cycle 2, Day 28 (< Median Cutpoint, n=15) | 8.0 [4.41 to 24.47]
  Cycle 2, Day 28 (> = Median Cutpoint, n=15) | 14.8 [13.26 to 22.89]
  Cycle 3, Day 1 (< Median Cutpoint, n=10) | 10.2 [5.20 to 14.84]
  Cycle 3, Day 1 (> = Median Cutpoint, n=10) | 15.8 [13.26 to 22.89]
  Cycle 3, Day 28 (< Median Cutpoint, n=6) | 14.2 [12.66 to 14.84]
  Cycle 5, Day 28 (< Median Cutpoint, n=2) | 14.2 [13.65 to 14.84]
  Cycle 5, Day 28 (> = Median Cutpoint, n=2) | 16.6 [12.66 to 20.53]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.4269, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.72 to 2.21] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.9290, Log Rank; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.51 to 1.86] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.8195, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.44 to 1.91] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.2210, Log Rank; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.26 to 1.38] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.4297, Log Rank; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.24 to 1.85] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.0522, Log Rank; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.06 to 1.11] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 7: Comparison: Sunitinib; Cycle 5, Day 28; Test type: Superiority or Other; p = 0.6949, Log Rank; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.05 to 7.00] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

33. Secondary Outcome: Comparison of Kaplan-Meier OS Curves After Stratification by < or > = Median Levels of Soluble E-Selectin at Baseline and Changes From Baseline
Description: OS=time from start of study treatment to death due to any cause. OS (in months) calculated as (date of death minus date of sunitinib first dose +1) divided by 30.4. For subjects not expiring their survival times were censored at last date of known contact they were known to be alive. Subjects lacking data beyond day of first dose of sunitinib had their survival time censored at Day 1 of sunitinib treatment. Groups are defined by < or > = median levels of soluble E-selectin at Baseline and after stratification by < or > = median changes from Baseline in soluble E-selectin at each time point.
Time Frame: Baseline to Cycle 1 (Day 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 4 (Day 28), Cycle 5 (Day 28) of Part 2
Population: MITT. n=number of subjects with soluble protein biomarkers at baseline and at the specified time point. At Cycle 3, Day 1 (< median cutpoint), Cycle 4, Day 28 (< median cutpoint, > = median cutpoint)and Cycle 5, Day 28 (< median cutpoint), median and/or CI were not able to be estimated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 53
months
  Cycle 1, Day 1 (< Median Cutpoint, n=26) | 6.5 [4.24 to 12.66]
  Cycle 1, Day 1 (> = Median Cutpoint, n=27) | 8.0 [4.51 to 13.65]
  Cycle 1, Day 28 (< Median Cutpoint, n=17) | 8.7 [4.57 to 24.47]
  Cycle 1, Day 28 (> = Median Cutpoint, n=17) | 6.5 [3.95 to 14.84]
  Cycle 2, Day 1 (< Median Cutpoint, n=14) | 11.2 [4.51 to 24.47]
  Cycle 2, Day 1 (> = Median Cutpoint, n=15) | 8.5 [5.23 to 13.26]
  Cycle 2, Day 28 (< Median Cutpoint, n=11) | 8.0 [4.41 to 24.47]
  Cycle 2, Day 28 (> = Median Cutpoint, n=11) | 14.8 [12.66 to 22.89]
  Cycle 3, Day 1 (> = Median Cutpoint, n=8) | 12.7 [5.07 to 14.84]
  Cycle 3, Day 28 (> = Median Cutpoint, n=4) | 15.3 [12.66 to 22.89]
  Cycle 5, Day 28 (> = Median Cutpoint, n=2) | 13.8 [12.66 to 14.84]
Statistical Analysis 1: Comparison: Sunitinib; Cycle 1, Day 1; Test type: Superiority or Other; p = 0.7660, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.51 to 1.65] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 2: Comparison: Sunitinib; Cycle 1, Day 28; Test type: Superiority or Other; p = 0.2682, Log Rank; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [0.72 to 3.23] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 3: Comparison: Sunitinib; Cycle 2, Day 1; Test type: Superiority or Other; p = 0.2726, Log Rank; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [0.69 to 3.70] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 4: Comparison: Sunitinib; Cycle 2, Day 28; Test type: Superiority or Other; p = 0.2787, Log Rank; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.22 to 1.55] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 5: Comparison: Sunitinib; Cycle 3, Day 1; Test type: Superiority or Other; p = 0.0241, Log Rank; Hazard Ratio (HR) = 4.4, 95% CI 2-sided [1.09 to 17.56] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 6: Comparison: Sunitinib; Cycle 3, Day 28; Test type: Superiority or Other; p = 0.0943, Log Rank; Hazard Ratio (HR) = 5.4, 95% CI 2-sided [0.59 to 48.81] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group
Statistical Analysis 7: Comparison: Sunitinib; Cycle 5, Day 28; Test type: Superiority or Other; p = 0.8084, Log Rank; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.04 to 11.79] — HR was based upon the ratio of > = median cutpoint group hazard to < median cutpoint group

34. Secondary Outcome: Immunohistochemical Staining of Paraffin Embedded Tumor Tissue
Description: Previously collected tumor paraffin block (or 12-20 10-micron slides prepared for the paraffin block) for correlative laboratory analysis.
Time Frame: Screening
Population: Samples were collected and stained from a subset of subjects. Due to the small sample size, no correlative analyses with clinical outcome were conducted.
Measure: Number; unit: samples
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 0

35. Secondary Outcome: Correlation of Polymorphisms in c-Kit, Flt-3 and c-Fms to Safety of Sunitinib
Description: A blood sample (6 mL) was collected and used to isolate DNA. These samples were not anonymized.
Time Frame: Within 7 days of Day 1
Population: c-Kit, Flt-3 and c-Fms to safety of Sunitinib samples were collected and analyzed. However, there was no statistics performed since power was insufficient.
Measure: Number; unit: pg/mL
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 0

36. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQOL) and Lung Cancer Related Symptoms as Assessed With the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30 scales: global health/QoL, functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much, global/QOL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms. Change: score at each visit in Part 2 minus baseline score in Part 1.
Time Frame: Baseline (Part 1) to Cycle1 (Days 1 [baseline], 28), Cycles 2 and 3 (Days 1, 28), and Cycle 4 (Day 1) in Part 2
Population: ITT. Number of participants analyzed = number of subjects with EORTC response (defined as having at least 1 item response on the EORTC). n=number of subjects with EORTC scale score at baseline and each specified time point. Data in cycles with less than 9 subjects are not reported due to lack of statistical reliability.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
scores on a scale
  Cycle 1, Day 1 Global Health Status /QoL (n=54) | -1.54 (3.580)
  Cycle 1, Day 28 Global Health Status /QoL (n=42) | -9.13 (3.964)
  Cycle 2, Day 1 Global Health Status /QoL (n=35) | -2.62 (3.361)
  Cycle 2, Day 28 Global Health Status /QoL (n=21) | -9.13 (4.704)
  Cycle 3, Day 1 Global Health Status /QoL (n=14) | 0.60 (7.175)
  Cycle 3, Day 28 Global Health Status /QoL (n=10) | -2.50 (8.056)
  Cycle 4, Day 1 Global Health Status /QoL (n=10) | 7.50 (4.883)
  Cycle 1, Day 1 Physical Functioning (n=54) | -6.79 (2.806)
  Cycle 1, Day 28 Physical Functioning (n=42) | -9.68 (2.363)
  Cycle 2, Day 1 Physical Functioning (n=35) | -7.43 (2.941)
  Cycle 2, Day 28 Physical Functioning (n=22) | -12.42 (4.771)
  Cycle 3, Day 1 Physical Functioning (n=15) | -5.78 (3.178)
  Cycle 3, Day 28 Physical Functioning (n=10) | -9.33 (7.647)
  Cycle 4, Day 1 Physical Functioning (n=10) | -2.00 (5.072)
  Cycle 1, Day 1 Role Functioning (n=54) | -16.05 (4.641)
  Cycle 1, Day 28 Role Functioning (n=42) | -20.63 (5.383)
  Cycle 2, Day 1 Role Functioning (n=35) | -13.81 (4.950)
  Cycle 2, Day 28 Role Functioning (n=22) | -28.03 (8.234)
  Cycle 3, Day 1 Role Functioning (n=15) | -16.67 (7.968)
  Cycle 3, Day 28 Role Functioning (n=10) | -15.00 (13.017)
  Cycle 4, Day 1 Role Functioning (n=10) | 8.33 (11.180)
  Cycle 1, Day 1 Emotional Functioning (n=54) | -2.16 (3.512)
  Cycle 1, Day 28 Emotional Functioning (n=42) | 3.57 (3.139)
  Cycle 2, Day 1 Emotional Functioning (n=35) | 1.90 (3.649)
  Cycle 2, Day 28 Emotional Functioning (n=21) | 1.98 (4.668)
  Cycle 3, Day 1 Emotional Functioning (n=14) | 13.10 (3.571)
  Cycle 3, Day 28 Emotional Functioning (n=10) | 12.50 (4.348)
  Cycle 4, Day 1 Emotional Functioning (n=10) | 24.17 (5.038)
  Cycle 1, Day 1 Cognitive Functioning (n=54) | -8.95 (3.138)
  Cycle 1, Day 28 Cognitive Functioning (n=42) | -3.57 (3.704)
  Cycle 2, Day 1 Cognitive Functioning (n=35) | -10.00 (3.817)
  Cycle 2, Day 28 Cognitive Functioning (n=21) | -10.32 (5.573)
  Cycle 3, Day 1 Cognitive Functioning (n=14) | 1.19 (3.692)
  Cycle 3, Day 28 Cognitive Functioning (n=10) | -1.67 (4.615)
  Cycle 4, Day 1 Cognitive Functioning (n=10) | 5.00 (5.000)
  Cycle 1, Day 1 Social Functioning (n=53) | -11.64 (4.250)
  Cycle 1, Day 28 Social Functioning (n=41) | -10.98 (5.417)
  Cycle 2, Day 1 Social Functioning (n=34) | -9.31 (5.228)
  Cycle 2, Day 28 Social Functioning (n=20) | -25.00 (7.204)
  Cycle 3, Day 1 Social Functioning (n=14) | -7.14 (5.980)
  Cycle 3, Day 28 Social Functioning (n=10) | -8.33 (11.453)
  Cycle 4, Day 1 Social Functioning (n=10) | 1.67 (7.222)
  Cycle 1, Day 1 Fatigue (n=54) | 13.48 (3.411)
  Cycle 1, Day 28 Fatigue (n=42) | 16.40 (3.921)
  Cycle 2, Day 1 Fatigue (n=35) | 8.25 (4.083)
  Cycle 2, Day 28 Fatigue (n=22) | 19.70 (6.025)
  Cycle 3, Day 1 Fatigue (n=15) | 8.15 (6.548)
  Cycle 3, Day 28 Fatigue (n=10) | 22.22 (11.355)
  Cycle 4, Day 1 Fatigue (n=10) | -1.11 (7.490)
  Cycle 1, Day 1 Nausea and Vomiting (n=54) | 5.56 (2.988)
  Cycle 1, Day 28 Nausea and Vomiting (n=42) | 11.90 (3.822)
  Cycle 2, Day 1 Nausea and Vomiting (n=35) | 6.67 (4.491)
  Cycle 2, Day 28 Nausea and Vomiting (n=22) | 6.82 (4.608)
  Cycle 3, Day 1 Nausea and Vomiting (n=15) | 5.56 (5.789)
  Cycle 3, Day 28 Nausea and Vomiting (n=10) | 11.67 (7.049)
  Cycle 4, Day 1 Nausea and Vomiting (n=10) | 1.67 (6.310)
  Cycle 1, Day 1 Pain (n=54) | 3.09 (4.228)
  Cycle 1, Day 28 Pain (n=42) | -0.79 (3.766)
  Cycle 2, Day 1 Pain (n=35) | 5.24 (4.572)
  Cycle 2, Day 28 Pain (n=22) | 0.76 (5.748)
  Cycle 3, Day 1 Pain (n=15) | 5.56 (6.640)
  Cycle 3, Day 28 Pain (n=10) | -1.67 (8.767)
  Cycle 4, Day 1 Pain (n=10) | -3.33 (7.778)
  Cycle 1, Day 1 Dyspnea (n=54) | 2.47 (3.396)
  Cycle 1, Day 28 Dyspnea (n=42) | 1.59 (3.760)
  Cycle 2, Day 1 Dyspnea (n=35) | -4.76 (4.352)
  Cycle 2, Day 28 Dyspnea (n=22) | -13.64 (6.454)
  Cycle 3, Day 1 Dyspnea (n=15) | -8.89 (3.940)
  Cycle 3, Day 28 Dyspnea (n=10) | 0.00 (8.607)
  Cycle 4, Day 1 Dyspnea (n=10) | -13.33 (7.370)
  Cycle 1, Day 1 Insomnia (n=54) | -3.09 (5.006)
  Cycle 1, Day 28 Insomnia (n=42) | -5.56 (5.671)
  Cycle 2, Day 1 Insomnia (n=35) | -2.86 (5.529)
  Cycle 2, Day 28 Insomnia (n=22) | 6.06 (8.672)
  Cycle 3, Day 1 Insomnia (n=15) | -2.22 (6.057)
  Cycle 3, Day 28 Insomnia (n=10) | 6.67 (10.887)
  Cycle 4, Day 1 Insomnia (n=10) | -20.00 (7.370)
  Cycle 1, Day 1 Appetite Loss (n=54) | 11.11 (5.138)
  Cycle 1, Day 28 Appetite Loss (n=42) | 20.63 (5.898)
  Cycle 2, Day 1 Appetite Loss (n=35) | 13.33 (7.633)
  Cycle 2, Day 28 Appetite Loss (n=22) | 10.61 (7.068)
  Cycle 3, Day 1 Appetite Loss (n=15) | 2.22 (7.606)
  Cycle 3, Day 28 Appetite Loss (n=10) | 13.3 (12.373)
  Cycle 4, Day 1 Appetite Loss (n=10) | -6.67 (10.887)
  Cycle 1, Day 1 Constipation (n=54) | 5.56 (4.109)
  Cycle 1, Day 28 Constipation (n=42) | -0.79 (5.266)
  Cycle 2, Day 1 Constipation (n=35) | 13.33 (4.965)
  Cycle 2, Day 28 Constipation (n=22) | -4.55 (6.317)
  Cycle 3, Day 1 Constipation (n=15) | -4.44 (6.397)
  Cycle 3, Day 28 Constipation (n=10) | -6.67 (6.667)
  Cycle 4, Day 1 Constipation (n=10) | -10.00 (5.092)
  Cycle 1, Day 1 Diarrhea (n=54) | -3.09 (2.206)
  Cycle 1, Day 28 Diarrhea (n=41) | 13.01 (5.058)
  Cycle 2, Day 1 Diarrhea (n=35) | 11.43 (4.916)
  Cycle 2, Day 28 Diarrhea (n=21) | 7.94 (5.589)
  Cycle 3, Day 1 Diarrhea (n=14) | 16.67 (6.767)
  Cycle 3, Day 28 Diarrhea (n=10) | 26.67 (9.686)
  Cycle 4, Day 1 Diarrhea (n=10) | 0.00 (9.938)
  Cycle 1, Day 1 Financial Difficulties (n=54) | 5.56 (2.607)
  Cycle 1, Day 28 Financial Difficulties (n=42) | 2.38 (2.381)
  Cycle 2, Day 1 Financial Difficulties (n=34) | 5.88 (4.331)
  Cycle 2, Day 28 Financial Difficulties (n=21) | 6.35 (5.453)
  Cycle 3, Day 1 Financial Difficulties (n=14) | 11.90 (7.500)
  Cycle 3, Day 28 Financial Difficulties (n=10) | 13.33 (10.184)
  Cycle 4, Day 1 Financial Difficulties (n=10) | 13.33 (10.184)

37. Secondary Outcome: Change From Baseline in HRQOL and Lung Cancer Related Symptoms as Assessed With the EORTC QLQ Lung Cancer Module (QLQ-LC13)
Description: QLQ-LC13 assessed lung cancer symptoms (dyspnea, coughing, dysphasia, hemoptysis, sore mouth, peripheral neuropathy, alopecia, chest pain, arm pain, shoulder pain, and pain in other parts). Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms. Change: score at each visit in Part 2 minus baseline score in Part 1.
Time Frame: Baseline (Part 1) to Cycle1 (Days 1 [baseline], 28), Cycles 2 and 3 (Days 1, 28), and Cycle 4 (Day 1) in Part 2
Population: as for outcome 36
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | First Carboplatin Plus Paclitaxel, Then Sunitinib
Number analyzed (Participants) | 84
scores on a scale
  Cycle 1, Day 1 Dyspnea (n=49) | 3.40 (3.008)
  Cycle 1, Day 28 Dyspnea (n=37) | 4.80 (3.030)
  Cycle 2, Day 1 Dyspnea (n=31) | 4.30 (4.112)
  Cycle 2, Day 28 Dyspnea (n=21) | 1.59 (4.490)
  Cycle 3, Day 1 Dyspnea (n=14) | -1.59 (3.466)
  Cycle 3, Day 28 Dyspnea (n=9) | 4.94 (6.705)
  Cycle 4, Day 1 Dyspnea (n=9) | 0.00 (3.208)
  Cycle 1, Day 1 Coughing (n=53) | -14.47 (5.120)
  Cycle 1, Day 28 Coughing (n=40) | -14.17 (5.048)
  Cycle 2, Day 1 Coughing (n=34) | -12.75 (5.077)
  Cycle 2, Day 28 Coughing (n=21) | -15.87 (7.496)
  Cycle 3, Day 1 Coughing (n=14) | -9.52 (5.445)
  Cycle 3, Day 28 Coughing (n=10) | -13.33 (7.370)
  Cycle 4, Day 1 Coughing (n=9) | -11.11 (7.857)
  Cycle 1, Day 1 Hemoptysis (n=53) | 0.63 (1.678)
  Cycle 1, Day 28 Hemoptysis (n=39) | 5.13 (3.362)
  Cycle 2, Day 1 Hemoptysis (n=33) | 2.02 (1.406)
  Cycle 2, Day 28 Hemoptysis (n=21) | -1.59 (2.795)
  Cycle 3, Day 1 Hemoptysis (n=14) | -2.38 (2.381)
  Cycle 3, Day 28 Hemoptysis (n=10) | 0.00 (0.000)
  Cycle 4, Day 1 Hemoptysis (n=9) | -3.70 (3.704)
  Cycle 1, Day 1 Sore Mouth (n=53) | -5.66 (3.782)
  Cycle 1, Day 28 Sore Mouth (n=40) | 20.00 (7.141)
  Cycle 2, Day 1 Sore Mouth (n=34) | 9.80 (7.111)
  Cycle 2, Day 28 Sore Mouth (n=21) | 12.70 (6.289)
  Cycle 3, Day 1 Sore Mouth (n=14) | 0.00 (3.494)
  Cycle 3, Day 28 Sore Mouth (n=10) | 10.00 (13.194)
  Cycle 4, Day 1 Sore Mouth (n=9) | -11.11 (7.857)
  Cycle 1, Day 1 Dysphasia (n=53) | -0.63 (3.298)
  Cycle 1, Day 28 Dysphasia (n=40) | 7.50 (4.697)
  Cycle 2, Day 1 Dysphasia (n=34) | 2.94 (5.145)
  Cycle 2, Day 28 Dysphasia (n=21) | -1.59 (2.795)
  Cycle 3, Day 1 Dysphasia (n=14) | -4.76 (4.762)
  Cycle 3, Day 28 Dysphasia (n=10) | -10.00 (5.092)
  Cycle 4, Day 1 Dysphasia (n=9) | -11.11 (5.556)
  Cycle 1, Day 1 Peripheral Neuropathy (n=53) | 42.14 (5.012)
  Cycle 1, Day 28 Peripheral Neuropathy (n=40) | 32.50 (5.402)
  Cycle 2, Day 1 Peripheral Neuropathy (n=34) | 28.43 (5.825)
  Cycle 2, Day 28 Peripheral Neuropathy (n=21) | 26.98 (7.841)
  Cycle 3, Day 1 Peripheral Neuropathy (n=14) | 23.81 (10.145)
  Cycle 3, Day 28 Peripheral Neuropathy (n=10) | 20.00 (10.184)
  Cycle 4, Day 1 Peripheral Neuropathy (n=9) | 7.41 (7.407)
  Cycle 1, Day 1 Alopecia (n=53) | 63.52 (5.407)
  Cycle 1, Day 28 Alopecia (n=40) | 40.83 (7.009)
  Cycle 2, Day 1 Alopecia (n=34) | 30.39 (7.627)
  Cycle 2, Day 28 Alopecia (n=20) | 11.67 (7.752)
  Cycle 3, Day 1 Alopecia (n=14) | 0.00 (0.000)
  Cycle 3, Day 28 Alopecia (n=10) | 0.00 (0.000)
  Cycle 4, Day 1 Alopecia (n=9) | 0.00 (0.000)
  Cycle 1, Day 1 Pain in Chest (n=53) | -8.18 (3.581)
  Cycle 1, Day 28 Pain in Chest (n=40) | -4.17 (3.415)
  Cycle 2, Day 1 Pain in Chest (n=34) | -0.98 (3.850)
  Cycle 2, Day 28 Pain in Chest (n=21) | 0.00 (3.984)
  Cycle 3, Day 1 Pain in Chest (n=14) | 4.76 (5.906)
  Cycle 3, Day 28 Pain in Chest (n=10) | 0.00 (7.027)
  Cycle 4, Day 1 Pain in Chest (n=9) | 7.41 (9.259)
  Cycle 1, Day 1 Pain in Arm or Shoulder (n=51) | -1.31 (4.171)
  Cycle 1, Day 28 Pain in Arm or Shoulder (n=39) | 0.85 (4.497)
  Cycle 2, Day 1 Pain in Arm or Shoulder (n=34) | 3.92 (6.257)
  Cycle 2, Day 28 Pain in Arm or Shoulder (n=21) | 3.17 (4.545)
  Cycle 3, Day 1 Pain in Arm or Shoulder (n=14) | 2.38 (4.228)
  Cycle 3, Day 28 Pain in Arm or Shoulder (n=10) | -6.67 (11.967)
  Cycle 4, Day 1 Pain in Arm or Shoulder (n=9) | -11.11 (11.111)
  Cycle 1, Day 1 Pain in Other Parts (n=47) | 3.55 (6.431)
  Cycle 1, Day 28 Pain in Other Parts (n=35) | -6.67 (5.925)
  Cycle 2, Day 1 Pain in Other Parts (n=27) | 12.35 (7.368)
  Cycle 2, Day 28 Pain in Other Parts (n=17) | 13.73 (8.603)
  Cycle 3, Day 1 Pain in Other Parts (n=14) | 11.90 (8.274)
  Cycle 3, Day 28 Pain in Other Parts (n=9) | -11.11 (9.623)
  Cycle 4, Day 1 Pain in Other Parts (n=9) | 0.00 (9.623)

ADVERSE EVENTS:
Description: Part 1 = adverse events (AEs) reported occurred during chemotherapy treatment. Part 2 = AEs reported occurred on or after the first dose of sunitinib.
Arm/Group | Carboplatin Plus Paclitaxel 172-225 mg/m2 (Part 1) | Sunitinib 50 mg (Part 2)
Serious Adverse Events (participants affected / at risk) | 29/84 | 29/66
Other Adverse Events (participants affected / at risk) | 82/84 | 60/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin Plus Paclitaxel 172-225 mg/m2 (Part 1) (N=84) | Sunitinib 50 mg (Part 2) (N=66)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 4 | 2
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 3
Disease progression (General disorders) | 1 | 7
Extravasation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 3
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Cardiac failure (Cardiac disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Coagulation time prolonged (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin Plus Paclitaxel 172-225 mg/m2 (Part 1) (N=84) | Sunitinib 50 mg (Part 2) (N=66)
Anaemia (Blood and lymphatic system disorders) | 28 | 12
Neutropenia (Blood and lymphatic system disorders) | 20 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 13
Constipation (Gastrointestinal disorders) | 23 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 24
Nausea (Gastrointestinal disorders) | 36 | 21
Vomiting (Gastrointestinal disorders) | 21 | 12
Asthenia (General disorders) | 14 | 17
Chest pain (General disorders) | 6 | 6
Chills (General disorders) | 6 | 7
Fatigue (General disorders) | 27 | 21
Mucosal inflammation (General disorders) | 6 | 8
Oedema peripheral (General disorders) | 12 | 7
Pain (General disorders) | 5 | 2
Pyrexia (General disorders) | 17 | 9
Weight decreased (Investigations) | 10 | 4
Anorexia (Metabolism and nutrition disorders) | 10 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 4
Dysgeusia (Nervous system disorders) | 5 | 10
Hypoaesthesia (Nervous system disorders) | 6 | 2
Neuropathy peripheral (Nervous system disorders) | 24 | 6
Paraesthesia (Nervous system disorders) | 8 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 9
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 0 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 4
Hypertension (Vascular disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.